CLINICAL TRIAL: NCT05928286
Title: Observational Study of Efficiency of the Drug Remaxol® (Inosine + Meglumine + Methionine + Nicotinamide + Succinic Acid) Used in the Treatment of Patients With Gallstone Disease Complicated With Obstructive Jaundice
Brief Title: Remaxol® Used in the Treatment of Patients With Gallstone Disease Complicated With Obstructive Jaundice
Status: Recruiting | Type: Observational
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: Remaxol\2022\02
Record Dates: First submitted 2022-12-28; First posted 2023-07-03 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-11

CONDITIONS: Gallstone Disease; Obstructive Jaundice
Keywords: Gallstone disease; Obstructive jaundice; Remaxol
MeSH Terms: conditions — Cholelithiasis; Jaundice, Obstructive | interventions — Remaxol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The test group: Standard therapy + Remaxol
  Interventions: Drug: Remaxol
- The control group: Standard therapy

INTERVENTIONS:
Drug: Remaxol — The perioperative infusion of Remaxol® (Inosine + Meglumine + Methionine + Nicotinamide + Succinic acid)
  Groups: The test group

SUMMARY:
Obstructive jaundice is observed in 10-80 % of gallstone disease cases. The conventional tactics for the management of patients with obstructive jaundice is to remove biliary hypertension by using endoscopic or minimally invasive methods. The final surgical treatment is performed after jaundice reduction and normalization of hepatic functions. We suppose that the administration of the drug Remaxol (Inosine + Meglumine + Methionine + Nicotinamide + Succinic acid) during the perioperative period shortens jaundice duration and decreases the complications rate.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Age from 18 to 70 years
3. Diagnosis: Gallstone disease. Cholelithiasis, choledocholithiasis. Obstructive jaundice.
4. Total bilirubin level in the blood in the range from 102.5 to 246 µmol/l.
5. Jaundice duration according to the patient is not more than 7 days.
6. Scheduled two-staged surgical treatment: 1) common bile duct decompression (endoscopic papillosphincterotomy and endoscopic lithoextraction); 2) laparoscopic cholecystectomy.

Exclusion Criteria:

1. Presence of other pathology causing jaundice syndrome (tumors, constrictions, etc.).
2. Acute cholangitis. Acute cholecystitis. Acute pancreatitis.
3. History of chronic viral hepatitis, hepatic cirrhosis.
4. Other surgical pathology aggravating the condition and/or requiring treatment.
5. Use in the treatment of drugs containing ademethionine.
6. CHF, functional class III-IV according to NYHA.
7. History of chronic kidney disease and/or creatinine level of more than 130 µmol/l.
8. Respiratory failure.
9. Impairment of consciousness.
10. Diabetes mellitus.
11. Psychic diseases.
12. Autoimmune diseases.
13. Tuberculosis, HIV infection.
14. Pregnancy, lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gallstone disease and obstructive jaundice, hospitalized for surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 286 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Therapy response rate: decrease of total bilirubin level down to 20.5 µmol/l Visit 3 or decrease in total bilirubin by 70% compared to Visit 1. | Up to 2 weeks
  Decrease of total bilirubin level down to 20.5 µmol/l Visit 3 or decrease in total bilirubin by 70% compared to Visit 1.

SECONDARY OUTCOMES:
Therapy response rate: decrease of total bilirubin level down to 61.5 µmol/l and lower by the time of cholecystectomy | Up to 2 weeks
  Decrease of total bilirubin level down to 61.5 µmol/l and lower by the time of cholecystectomy, after successful common bile duct decompression.
Complication rate in the postoperative period | Up to 2 weeks
  Acute pancreatitis, acute renal failure, acute heart failure, pneumonia, stress hyperglycemia, infectious complications
Total hospitalization duration in days (in case of two-staged surgical treatment). | Up to 2 weeks
  Total hospitalization duration in days
Total hyperbilirubinemia duration (in days) after the beginning of fluid administration. | Up to 2 weeks
  Total hyperbilirubinemia duration (in days) after the beginning of fluid administration
Interval (in days) between surgical interventions | Up to 2 weeks
  Interval (in days) between surgical interventions
Change of hepatic function tests (AST,) | Baseline, on the day after surgery, up to 2 weeks
  Change of hepatic function tests (AST) relative to baseline values, on the day after common bile duct decompression, by the time of cholecystectomy, on the day after cholecystectomy, and on the day of hospitalization termination.
Change of hepatic function tests ( ALT) | Baseline, on the day after surgery, up to 2 weeks
  Change of hepatic function tests (ALT) relative to baseline values, on the day after common bile duct decompression, by the time of cholecystectomy, on the day after cholecystectomy, and on the day of hospitalization termination.
Change of hepatic function test ( AP) | Baseline, on the day after surgery, up to 2 weeks
  Change of hepatic function test ( AP) relative to baseline values, on the day after common bile duct decompression, by the time of cholecystectomy, on the day after cholecystectomy, and on the day of hospitalization termination.
Change of hepatic function test (GGTP) | Baseline, on the day after surgery, up to 2 weeks
  Change of hepatic function test (GGTP) relative to baseline values, on the day after common bile duct decompression, by the time of cholecystectomy, on the day after cholecystectomy, and on the day of hospitalization termination.
Change of hepatic function tests (protein, albumin, fibrinogen) | Baseline, on the day after surgery, up to 2 weeks
  Change of hepatic function tests (protein, albumin, fibrinogen) relative to baseline values, on the day after common bile duct decompression, by the time of cholecystectomy, on the day after cholecystectomy, and on the day of hospitalization termination.
Change of PTI | Baseline, on the day after surgery, up to 2 weeks
  Change of PTI relative to baseline values, on the day after common bile duct decompression, by the time of cholecystectomy, on the day after cholecystectomy, and on the day of hospitalization termination.
Change of renal function test (urea) | Baseline, on the day after surgery, up to 2 weeks
  Change of renal function test (urea) relative to baseline values, on the day after common bile duct decompression, by the time of cholecystectomy, on the day after cholecystectomy, and on the day of hospitalization termination.
Change of renal function test (creatinine) | Baseline, on the day after surgery, up to 2 weeks
  Change of renal function test (creatinine) relative to baseline values, on the day after common bile duct decompression, by the time of cholecystectomy, on the day after cholecystectomy, and on the day of hospitalization termination.
Number of patients whose cholecystectomy was delayed till next hospitalization because of the insufficient dynamics of decrease in bilirubinemia. | Up to 2 weeks
  Number of patients whose cholecystectomy was delayed till next hospitalization because of the insufficient dynamics of decrease in bilirubinemia.

CONTACTS AND LOCATIONS:
Locations (9):
- Russia (9):
  - Krai Clinical Hospital, Barnaul
  - Hospital for War Veterans, Kazan'
  - City Clinical Hospital No. 7, Nizhny Novgorod
  - Pavlov Ryazan State Medical University, Ryazan
  - Dzhanelidze St. Petersburg Research Institute of Emergency Medicine, Saint Petersburg
  - St. Elizabeth Hospital, Saint Petersburg
  - Samara State Medical University, Samara
  - Mirotvortsev University Clinical Hospital No. 1, Saratov
  - Kuvatov Republican Clinical Hospital, Ufa

IPD SHARING:
Plan to Share IPD: No